CLINICAL TRIAL: NCT06865651
Title: A 12-week Randomized, Participant and Investigator-blinded, Placebo-controlled, Exploratory Study in Adult Participants With Chronic Urticaria to Assess the Efficacy and Safety and Explore the Mechanism of Action of Remibrutinib (LOU064)
Brief Title: Study of Remibrutinib (LOU064) Efficacy and Safety and Exploration of Its Mechanism of Action in Participants With Chronic Urticaria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CLOU064M12101
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Urticaria (CU): Chronic Inducible Urticaria (CINDU) and Chronic Spontaneous Urticaria (CSU)
Keywords: Remibrutinib; LOU064; Chronic urticaria; CINDU; CSU; Symptomatic dermographism; Cold urticaria; Cholinergic urticaria; Heat urticaria; Solar urticaria; Delayed pressure urticaria; Aquagenic urticaria; Contact urticaria
MeSH Terms: conditions — Chronic Urticaria; Chronic Inducible Urticaria; Familial dermographism; Cold Urticaria; Urticaria, Solar | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LOU064-CINDU (Experimental): Diagnosis of Chronic Inducible Urticaria (CINDU), symptoms of symptomatic dermographism urticaria, cold urticaria, cholinergic urticaria, heat urticaria, solar urticaria, urticaria as diagnosed by pressure, evidence of urticaria after exposure to water, evidence of urticaria following contact to identified material causing urticaria symptoms.
  Interventions: Drug: Remibrutinib
- LOU064-CSU (Experimental): Diagnosis of Chronic Spontaneous Urticaria (CSU) not adequately controlled
  Interventions: Drug: Remibrutinib
- Placebo-CINDU (Placebo Comparator): Diagnosis of Chronic Inducible Urticaria (CINDU), symptoms of symptomatic dermographism urticaria, cold urticaria, cholinergic urticaria, heat urticaria, solar urticaria, urticaria as diagnosed by pressure, evidence of urticaria after exposure to water, evidence of urticaria following contact to identified material causing urticaria symptoms.
  Interventions: Drug: Placebo
- Placebo-CSU (Placebo Comparator): Diagnosis of Chronic Spontaneous Urticaria (CSU) not adequately controlled
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remibrutinib — tablets
  Other Names: LOU064
  Arms: LOU064-CINDU; LOU064-CSU
Drug: Placebo — tablets
  Arms: Placebo-CINDU; Placebo-CSU

SUMMARY:
The purpose of this study is to explore the effect and Mechanism of Action (MoA) of remibrutinib (LOU064) vs. placebo on clinical outcomes in participants with Chronic Urticaria (CU), including both Chronic Spontaneous Urticaria (CSU) and Chronic Inducible Urticaria (CINDU).

DETAILED DESCRIPTION:
This is a randomized, parallel-group, participant and investigator-blinded, placebo controlled, multi-center study in approximately 44 adult participants that are diagnosed with a form of CU and have symptoms despite treatment with H1-antihistamines. The following nine subtypes of CU are included:

* CINDU cohorts: Symptomatic dermographism, Cold urticaria, Cholinergic urticaria, Heat urticaria, Solar urticaria, Delayed pressure urticaria, Aquagenic urticaria, Contact urticaria
* CSU The study will attempt to enroll approximately 4-5 participants for each subtype. Participants will undergo a screening period for completion of the assessment to check eligibility criteria which will take approximately up to 4 weeks. After enrollment, the treatment will be initiated. Participants will either receive remibrutinib or placebo for 12 weeks. Participants have an end of study visit approximately 7 days after the last dose. All participants will have a safety follow-up phone call approximately 30 days after last treatment administration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male and female participants ≥ 18 years of age at the time of signing of the informed consent forms.
3. CINDU patients: Confirmed diagnosis of CINDU with a duration of ≥ 4 months (defined as onset of CINDU with supporting documentation (e.g. medical record, clinical history, photographs) and inadequate control with H1-AH at local label approved doses at the time of randomization. The response to the provocation test for each CINDU subtype is required before randomization (either during screening or prior to randomization on Day 1):
4. CINDU patients: Patients should be symptomatic for their most bothersome symptom as assessed with the USDD during baseline with a NRS score of 3 or more
5. CSU patients: Diagnosis of CSU (acc. to Zuberbier et al 2022c) not adequately controlled with H1-AH at approved doses alone for at least 4 weeks prior to randomization, as defined by all of the following:

   * UAS7 score (range 0-42) ≥ 16 and HSS7 (range 0-21) ≥ 8 during 7 days prior to randomization
   * CSU for ≥ 6 months
6. Participants must be willing and able to attend the protocol defined test procedure throughout the study.

Exclusion Criteria:

1. Participants who have a familial/hereditary form (e.g. familial cold autoinflammatory syndrome, familial cold urticaria) of the target CINDU that is being considered for the participant's inclusion in this study.
2. Diseases, other than CSU or CINDU, with urticaria or angioedema symptoms including but not limited to:

   * urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa),
   * food allergies yielding urticaria symptoms when the allergen is not avoided by the dietary habits of the participant
   * hereditary or acquired angioedema.
3. CINDU patients only: To prevent any confounding effect of CSU symptoms, the CINDU study population will consist of participants with predominant CINDU and should not have a significant share of CSU symptoms (that might make the assessment of CINDU symptoms difficult) as per the investigator's judgement.
4. CSU patients only: Patients should have no relevant inducible urticaria trigger
5. Any other skin disease associated with chronic itching that might influence, in the investigator's opinion, the study evaluations and results (e.g., atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.) or skin diseases associated with only wheals and no itch e.g asymptomatic dermographism
6. Known or suspected ongoing, chronic or recurrent infectious disease including but not limited to opportunistic infections (e.g., tuberculosis, atypical mycobacterioses, listeriosis or aspergillosis) and/or known positivity for Human Immunodeficiency Virus (HIV) infection.
7. Evidence of an ongoing Hepatitis C infection (defined by the detection at screening of Hepatitis C virus antibodies (anti-HCVAb) and hepatitis C ribonucleic acid (HCV-RNA) in participants who are positive for anti-HCVAb) and/or an ongoing Hepatitis B infection (defined by the detection of Hepatitis B virus surface antigen (HBsAg) and/or hepatitis B virus (HBV)-DNA at screening; participants who are positive for anti-hepatitis B core (HBc) antibodies but who are negative for antibodies against HBsAg and HBV-DNA can be included into the study if they agree to monitoring for HBsAg and HBV-DNA reactivation).
8. Major surgery within 8 weeks prior to screening or planned surgery for the duration of the study.
9. Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 12 months prior to Screening), neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant.
10. Uncontrolled disease states, such as asthma, or inflammatory bowel disease, or any other disease where flares are commonly treated with oral or parenteral corticosteroids.
11. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
12. History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or BUN values, or abnormal urinary constituents (e.g. proteinuria, hematuria)

    * Evidence of urinary obstruction, or difficulty in voiding at screening
    * Evidence of congenital renal abnormalities with known effect on renal function
    * Calculated eGFR < 60 mL/min
13. Hematology parameters at screening:

    * Hemoglobin: < 10 g/dL
    * Platelets: < 100,000/mm3
    * Leucocytes: < 3,000/mm3
    * Neutrophils:< 1,500/mm3
14. History or current hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis or hepatic failure or Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) levels of more than 1.5 x upper limit of normal (ULN) or International Normalized Ratio (INR) of more than 1.5 at screening
15. Use of other investigational drugs s within 5 half-lives or within 30 days (for small molecules) prior to Screening or until the expected pharmacodynamic (PD) effect has returned to baseline (for biologics), whichever is longer; or longer if required by local regulations
16. Contraindications to or hypersensitivity to remibrutinib (or its excipients or to drugs of similar chemical classes) or other substances provided to the subjects as rescue medication to control symptoms, such as antihistamines.
17. Participants taking prohibited therapies as listed in Section 6.6.2. In particular patients with pretreatment with remibrutinib or another BTK-inhibitor within 4 months prior to randomization.
18. History of live or live attenuated vaccine within 6 weeks prior to randomization or requirement to receive these vaccinations at any time during the study drug treatment.
19. Requirement for anti-platelet medication, except for acetylsalicylic acid up to 100 mg/d or clopidogrel up to 75 mg/d which are allowed. The use of dual anti-platelet therapy (e.g., acetylsalicylic acid + clopidogrel) is prohibited.
20. Requirement for anticoagulant medication (for example, warfarin or Novel Oral Anti-Coagulants (NOAC)).
21. History of gastrointestinal bleeding, e.g., in association with use of nonsteroidal anti-inflammatory drugs (NSAID), that was clinically relevant (e.g., where intervention was indicated or requiring hospitalization or blood transfusion)
22. Significant bleeding risk or coagulation disorders.
23. Known history or evidence of ongoing alcohol or drug abuse within the last 6 months before randomization as per source records.
24. Pregnant or nursing (breast feeding) women.
25. Women of child-bearing potential, defined as fertile, following menarche and until becoming post-menopausal unless they are permanent sterile or they are using highly effective methods of contraception during dosing for 7 days after stopping study treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Note that periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Bilateral oophorectomy with or without hysterectomy, total hysterectomy or bilateral salpingectomy at least six weeks prior to the first dose of study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered to be not of child-bearing potential.
    * Bilateral tubal occlusion, Bilateral tubal ligation (at least six weeks prior to the first dose of study treatment)
    * Male partner sterilization (vasectomy) of male partner(s) of the female participant at least six months prior to screening). The vasectomized male partner should be sole partner for that participant and received medical assessment of the surgical success.
    * Use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.

The decision on the contraceptive method should be reviewed at least every 3 months to evaluate the individual need and compatibility of the method chosen. In case of use of hormonal contraception, women should have been stable on the same method for a minimum of 3 months before taking study treatment. Women are considered post-menopausal if they have no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Women are considered not of child-bearing potential if they are post-menopausal or permanently sterileor have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral salpingectomy at least six weeks prior to first dose of study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child-bearing potential.

If local regulations are more stringent than the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-07 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in the weekly most bothersome symptom Numeric Rating Scale (NRS) score on the Urticaria Symptom Daily Diary (USDD) | Baseline, Week 6
  To investigate the efficacy of remibrutinib versus placebo for the most bothersome symptom in CINDU patients. The USDD was developed to assess daily exposure and avoidance of triggers, severity of urticaria symptoms (including NRS for pain itch and burning). On the first day of completion, the participants will be asked which symptom (itch, pain, and burning) is the most bothersome symptom of urticaria.
Absolute change from baseline in Urticaria Control Test 7 (UCT7) weekly scores | Baseline, Week 6
  To investigate the impact of remibrutinib versus placebo on urticaria symptom control. The UCT is a 4-item PRO measure developed to assess disease control in patients with CU specifically CINDU and CSU. It has a 7-day recall period and participants respond with how much they were bothered by their urticaria symptoms, what is the impact on QoL, how often the treatment did not control their urticaria and their overall perception of disease control. Each question can be scored on a scale from 0 to 4 and the overall score ranges from 0 (no control) to 16 (maximum control). The cut-off value for disease control was established at 12. Participants with a score above 12 are considered controlled. A minimally important difference of 3 points was validated as reflective of a clinically relevant change of control.

SECONDARY OUTCOMES:
Absolute change from baseline in Urticaria Control test 7 (UCT7) weekly scores | Baseline, Week 2 and Week 12
  To investigate the impact of remibrutinib versus placebo on urticaria symptom control and quality of life. The UCT is a 4-item PRO measure developed to assess disease control in patients with CU specifically CINDU and CSU. It has a 7-day recall period and participants respond with how much they were bothered by their urticaria symptoms, what is the impact on QoL, how often the treatment did not control their urticaria and their overall perception of disease control. Each question can be scored on a scale from 0 to 4 and the overall score ranges from 0 (no control) to 16 (maximum control). The cut-off value for disease control was established at 12. Participants with a score above 12 are considered controlled. A minimally important difference of 3 points was validated as reflective of a clinically relevant change of control.
Dermatology Life Quality Index (DLQI) response defined as DLQI= 0-1 | Week 2, Week 6 and Week 12
  To investigate the impact of remibrutinib versus placebo on urticaria symptom control and quality of life. The DLQI is a 10-item (grouped in 6 domains) dermatology-specific Quality of Life (QoL) measure. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse dermatology QoL). For DLQI, the domain scores are calculated for: Symptoms and Feelings (0-6), Daily Activities (0-6), Leisure (0-6), Work and School (0-3), Personal Relationships (0-6) and Treatment (0-3). A DLQI score of > 10 is relevant for a very large impact on patients' life and justification for a biologic prescription for example in psoriasis.
Absolute change from baseline in USDD weekly component scores; this includes the change in itch, pain and burning numeric rating scale (NRS) from baseline. | Baseline, Week 2, Week 6 and Week 12
  To investigate the change in symptoms in participants treated with remibrutinib versus placebo. The USDD was developed to assess daily exposure and avoidance of triggers, severity of urticaria symptoms (including NRS for pain itch and burning). On the first day of completion, the participants will be asked which symptom (itch, pain, and burning) is the most bothersome symptom of urticaria.
Number of Participants With Adverse Events of Special Interest (AESI) | 17 weeks
  To investigate the safety of remibrutinib versus placebo in patients with Chronic Urticaria

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Endeavor Health, Glenview, Illinois
- France (4):
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
- Germany (4):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Tübingen
- Poland (3):
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.